CLINICAL TRIAL: NCT03135067
Title: Secondary Distribution of HIV Self-tests: an Innovative Strategy for Promoting Partner Testing and Reducing HIV Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Impact Research & Development Organization (Other); RTI International (Other); University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 828100; R01MH111602 (NIH)
Record Dates: First submitted 2017-04-17; First posted 2017-05-01 (Actual); Results first posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV self-testing; female sex workers; partner testing; couples testing; transactional sex
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Female sex worker hotspots and beach communities in the Nyanza region of Kenya will be grouped into clusters that will be randomly assigned to receive the intervention (provision of multiple HIV self-test kits over time) or control (provision of clinic-based HIV testing referral vouchers over time). About 66 clusters, with an average of 30 participants per cluster, will be selected for the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Provision of multiple self-tests (Experimental): Participants in intervention clusters will be given multiple HIV self-test kits, testing instructions, and advice to use their discretion when offering self-tests to selected sexual partners. Participants will be encouraged to offer self-tests primarily to current and potential partners with whom unprotected sex is likely. All participants will be encouraged to use condoms with sexual partners. Participants will also be advised to assess the risk of intimate partner violence (IPV) as a result of offering self-tests to partners. Participants will have opportunities to obtain additional HIV self-test kits on a monthly basis.
  Interventions: Behavioral: Provision of multiple self-tests
- Referral vouchers for VCT (No Intervention): Participants will be given a multiple referral vouchers for HIV testing to distribute to their sexual partners. All participants will be encouraged to use condoms with sexual partners. These referral vouchers will encourage the partners to seek HIV counseling & testing services in local clinics. Participants will also be advised to assess the risk of intimate partner violence (IPV) as a result of offering referral vouchers to partners. Participants will have opportunities to obtain additional referral vouchers on a monthly basis.

INTERVENTIONS:
Behavioral: Provision of multiple self-tests — Participants will be given multiple Oraquick Advance HIV-1/2 test kits for testing themselves more frequently and for offering to selected sexual partners. The self-test kits will be given to participants on a monthly basis as needed. The intervention is designed to facilitate partner and couples testing, with resulting reduction in risky sexual behavior and HIV incidence among participants.
  Arms: Provision of multiple self-tests

SUMMARY:
This cluster randomized trial will assess whether the provision of multiple oral-fluid based HIV self-test kits to HIV-negative women at high risk of acquiring HIV in western Kenya is an approach that promotes HIV testing among women's sexual partners, facilitates better sexual decision making, and reduces women's risk of acquiring HIV.

DETAILED DESCRIPTION:
The study will recruit HIV-negative adult women who had two or more sexual partners within the past four weeks in the Nyanza region of Kenya. Beach communities and female sex worker hotspots will be randomized to an intervention group or a control group. In intervention clusters, participants will receive multiple oral fluid-based HIV test kits over a period of up to 24 months, training on how to use the tests, and encouragement to offer tests to current and potential sexual partners with whom sex without condoms is likely. In the comparison clusters, participants will be given referral vouchers for clinic-based HIV testing over a period of up to 24-months and encouraged to distribute these vouchers to sexual partners.

Data will be collected from study participants at baseline on demographic and socio-economic characteristics, self-reported sexual behavior, HIV testing history, intimate partner violence history, and mental health outcomes. Follow-up data collection will occur every 6 months. Each month, participants will be sent an invitation to participate in short mobile phone based text message surveys. HIV testing of participants will occur at baseline and at 6 monthly intervals.

Based on their reported use of the HIV self-tests, participants will be invited for qualitative interviews to learn more about their interactions with partners with regard to the distribution of self-tests and referral vouchers. Participants will also be given information to distribute to some of their male partners so that those partners can contact study staff to participate in qualitative interviews that will inquired about their perceptions of self-tests.

The study has 3 specific aims. Aim 1 will determine the intervention's effect on uptake of HIV testing and identification of HIV infection among participants' sexual partners, self-reported sexual behavior of participants with partners whose HIV status was HIV-positive or not known, and HIV incidence among participants. Aim 2 will use a mixed methods approach to assessing safety and perceptions of the intervention by participants and their sexual partners. Aim 3 will assess the cost-effectiveness of the intervention and obtain information necessary to inform scale-up of the intervention in Kenya and other countries.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Currently resides in the study area
* Has resided in the study area for at least 6 months in the year prior to enrollment
* Intends to stay in the study area for at least 24 months
* Reports two or more sexual partners within the past 4 weeks at time of screening
* HIV negative
* Ownership or access to a mobile phone
* Willing and able to provide informed consent

Exclusion Criteria:

* Younger than 18 years old
* Does not currently live in the study area or has not for 6 of the last 12 months, or does not plan to for at least the next 24 months
* Fewer than two sexual partners in the last four weeks at time of screening
* HIV positive
* Has no access to a mobile phone
* Enrolled in another HIV prevention study
* Cannot or will not provide informed consent

  * Males will self-select to participate by contacting the study staff using the information provided by willing index participants. There are no inclusion or exclusion criteria for the men who select to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2102 (Actual)
Dates: Start 2017-06-04 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Thirumurthy, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Impact Research and Development Organization, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Unaids, THE GAP REPORT. 2014: Geneva, Switzerland.
- [Background] Staveteig, S., et al., Demographic Patterns of HIV Testing Uptake in Sub-Saharan Africa. DHS Comparative Reports No. 30. Calverton, Maryland, USA: ICF International. 2013.
- [Background] Suthar AB, Ford N, Bachanas PJ, Wong VJ, Rajan JS, Saltzman AK, Ajose O, Fakoya AO, Granich RM, Negussie EK, Baggaley RC. Towards universal voluntary HIV testing and counselling: a systematic review and meta-analysis of community-based approaches. PLoS Med. 2013 Aug;10(8):e1001496. doi: 10.1371/journal.pmed.1001496. Epub 2013 Aug 13. PMID 23966838
- [Background] Sharma M, Ying R, Tarr G, Barnabas R. Systematic review and meta-analysis of community and facility-based HIV testing to address linkage to care gaps in sub-Saharan Africa. Nature. 2015 Dec 3;528(7580):S77-85. doi: 10.1038/nature16044. PMID 26633769
- [Background] Chamie G, Clark TD, Kabami J, Kadede K, Ssemmondo E, Steinfeld R, Lavoy G, Kwarisiima D, Sang N, Jain V, Thirumurthy H, Liegler T, Balzer LB, Petersen ML, Cohen CR, Bukusi EA, Kamya MR, Havlir DV, Charlebois ED. A hybrid mobile approach for population-wide HIV testing in rural east Africa: an observational study. Lancet HIV. 2016 Mar;3(3):e111-9. doi: 10.1016/S2352-3018(15)00251-9. Epub 2016 Jan 26. PMID 26939734
- [Background] National AIDS and STI Control Programme (NASCOP), K., Kenya AIDS Indicator Survey 2012: Final Report. 2014, NASCOP: Nairobi.
- [Background] National AIDS and STI Control Programme, Kenya AIDS Indicator Survey 2012: Nyanza Region Fact Sheet 2014, Nairobi, Kenya: NASCOP.
- [Background] Ng'ang'a A, Waruiru W, Ngare C, Ssempijja V, Gachuki T, Njoroge I, Oluoch P, Kimanga DO, Maina WK, Mpazanje R, Kim AA; KAIS Study Group. The status of HIV testing and counseling in Kenya: results from a nationally representative population-based survey. J Acquir Immune Defic Syndr. 2014 May 1;66 Suppl 1(Suppl 1):S27-36. doi: 10.1097/QAI.0000000000000102. PMID 24732818
- [Background] Baral S, Beyrer C, Muessig K, Poteat T, Wirtz AL, Decker MR, Sherman SG, Kerrigan D. Burden of HIV among female sex workers in low-income and middle-income countries: a systematic review and meta-analysis. Lancet Infect Dis. 2012 Jul;12(7):538-49. doi: 10.1016/S1473-3099(12)70066-X. Epub 2012 Mar 15. PMID 22424777
- [Background] WHO, Preventing HIV in Sex Work Settings in sub Saharan Africa. 2011, World Health Organization: Geneva.
- [Background] Beyrer C, Crago AL, Bekker LG, Butler J, Shannon K, Kerrigan D, Decker MR, Baral SD, Poteat T, Wirtz AL, Weir BW, Barre-Sinoussi F, Kazatchkine M, Sidibe M, Dehne KL, Boily MC, Strathdee SA. An action agenda for HIV and sex workers. Lancet. 2015 Jan 17;385(9964):287-301. doi: 10.1016/S0140-6736(14)60933-8. Epub 2014 Jul 22. PMID 25059950
- [Background] Vandenhoudt HM, Langat L, Menten J, Odongo F, Oswago S, Luttah G, Zeh C, Crucitti T, Laserson K, Vulule J, Buve A. Prevalence of HIV and other sexually transmitted infections among female sex workers in Kisumu, Western Kenya, 1997 and 2008. PLoS One. 2013;8(1):e54953. doi: 10.1371/journal.pone.0054953. Epub 2013 Jan 23. PMID 23372801
- [Background] Odek WO, Githuka GN, Avery L, Njoroge PK, Kasonde L, Gorgens M, Kimani J, Gelmon L, Gakii G, Isac S, Faran E, Musyoki H, Maina W, Blanchard JF, Moses S. Estimating the size of the female sex worker population in Kenya to inform HIV prevention programming. PLoS One. 2014 Mar 3;9(3):e89180. doi: 10.1371/journal.pone.0089180. eCollection 2014. PMID 24595029
- [Background] Kiwanuka N, Ssetaala A, Nalutaaya A, Mpendo J, Wambuzi M, Nanvubya A, Sigirenda S, Kitandwe PK, Nielsen LE, Balyegisawa A, Kaleebu P, Nalusiba J, Sewankambo NK. High incidence of HIV-1 infection in a general population of fishing communities around Lake Victoria, Uganda. PLoS One. 2014 May 27;9(5):e94932. doi: 10.1371/journal.pone.0094932. eCollection 2014. PMID 24866840
- [Background] Kwena Z, Mwanzo I, Shisanya C, Camlin C, Turan J, Achiro L, Bukusi E. Predictors of extra-marital partnerships among women married to fishermen along Lake Victoria in Kisumu County, Kenya. PLoS One. 2014 Apr 18;9(4):e95298. doi: 10.1371/journal.pone.0095298. eCollection 2014. PMID 24747951
- [Background] Camlin CS, Kwena ZA, Dworkin SL. Jaboya vs. jakambi: Status, negotiation, and HIV risks among female migrants in the "sex for fish" economy in Nyanza Province, Kenya. AIDS Educ Prev. 2013 Jun;25(3):216-31. doi: 10.1521/aeap.2013.25.3.216. PMID 23631716
- [Background] Choko AT, Desmond N, Webb EL, Chavula K, Napierala-Mavedzenge S, Gaydos CA, Makombe SD, Chunda T, Squire SB, French N, Mwapasa V, Corbett EL. The uptake and accuracy of oral kits for HIV self-testing in high HIV prevalence setting: a cross-sectional feasibility study in Blantyre, Malawi. PLoS Med. 2011 Oct;8(10):e1001102. doi: 10.1371/journal.pmed.1001102. Epub 2011 Oct 4. PMID 21990966
- [Background] Johnson C, Baggaley R, Forsythe S, van Rooyen H, Ford N, Napierala Mavedzenge S, Corbett E, Natarajan P, Taegtmeyer M. Realizing the potential for HIV self-testing. AIDS Behav. 2014 Jul;18 Suppl 4:S391-5. doi: 10.1007/s10461-014-0832-x. PMID 24986599
- [Background] Napierala Mavedzenge S, Baggaley R, Corbett EL. A review of self-testing for HIV: research and policy priorities in a new era of HIV prevention. Clin Infect Dis. 2013 Jul;57(1):126-38. doi: 10.1093/cid/cit156. Epub 2013 Mar 13. PMID 23487385
- [Background] Lee VJ, Tan SC, Earnest A, Seong PS, Tan HH, Leo YS. User acceptability and feasibility of self-testing with HIV rapid tests. J Acquir Immune Defic Syndr. 2007 Aug 1;45(4):449-53. doi: 10.1097/QAI.0b013e318095a3f3. PMID 17554213
- [Background] Carballo-Dieguez A, Frasca T, Balan I, Ibitoye M, Dolezal C. Use of a rapid HIV home test prevents HIV exposure in a high risk sample of men who have sex with men. AIDS Behav. 2012 Oct;16(7):1753-60. doi: 10.1007/s10461-012-0274-2. PMID 22893194
- [Background] Thirumurthy, H., et al. Acceptability and feasibility of a novel approach to promote HIV testing in sexual and social networks using HIV self-tests. . in International AIDS Society (IAS) conference. 2015. Vancouver, Canada.
- [Background] Choko AT, MacPherson P, Webb EL, Willey BA, Feasy H, Sambakunsi R, Mdolo A, Makombe SD, Desmond N, Hayes R, Maheswaran H, Corbett EL. Uptake, Accuracy, Safety, and Linkage into Care over Two Years of Promoting Annual Self-Testing for HIV in Blantyre, Malawi: A Community-Based Prospective Study. PLoS Med. 2015 Sep 8;12(9):e1001873. doi: 10.1371/journal.pmed.1001873. eCollection 2015 Sep. PMID 26348035
- [Background] Figueroa C, Johnson C, Verster A, Baggaley R. Attitudes and Acceptability on HIV Self-testing Among Key Populations: A Literature Review. AIDS Behav. 2015 Nov;19(11):1949-65. doi: 10.1007/s10461-015-1097-8. PMID 26054390
- [Background] Kalibala S, Tun W, Cherutich P, Nganga A, Oweya E, Oluoch P. Factors associated with acceptability of HIV self-testing among health care workers in Kenya. AIDS Behav. 2014 Jul;18 Suppl 4(Suppl 4):S405-14. doi: 10.1007/s10461-014-0830-z. PMID 24974123
- [Background] Kalibala, S., W. Tun, and W. Muraah, Feasibility and acceptability of HIV self testing among health care workers: results of a pilot programme in two hospitals in Kenya, in XVIII International AIDS Conference, Abstract WEPDC205, Editor. 2010: Vienna, Austria 18-23 July.
- [Background] Consolidated Guidelines on HIV Testing Services: 5Cs: Consent, Confidentiality, Counselling, Correct Results and Connection 2015. Geneva: World Health Organization; 2015 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK316021/ PMID 26378328
- [Background] National AIDS and STD Control Programme, Guidelines for HIV Testing and Counselling in Kenya, Ministry of Public Health and Sanitation Kenya, Editor. 2008, Nairobi: NASCOP.
- [Background] National AIDS and STI Control Programme, Guidelines for HIV Testing Services in Kenya. 2015, Nairobi: National AIDS Control Programme.
- [Background] Kimbrough LW, Fisher HE, Jones KT, Johnson W, Thadiparthi S, Dooley S. Accessing social networks with high rates of undiagnosed HIV infection: The social networks demonstration project. Am J Public Health. 2009 Jun;99(6):1093-9. doi: 10.2105/AJPH.2008.139329. Epub 2009 Apr 16. PMID 19372521
- [Background] Golden MR, Kerani RP, Stenger M, Hughes JP, Aubin M, Malinski C, Holmes KK. Uptake and population-level impact of expedited partner therapy (EPT) on Chlamydia trachomatis and Neisseria gonorrhoeae: the Washington State community-level randomized trial of EPT. PLoS Med. 2015 Jan 15;12(1):e1001777. doi: 10.1371/journal.pmed.1001777. eCollection 2015 Jan. PMID 25590331
- [Background] Balan IC, Carballo-Dieguez A, Frasca T, Dolezal C, Ibitoye M. The impact of rapid HIV home test use with sexual partners on subsequent sexual behavior among men who have sex with men. AIDS Behav. 2014 Feb;18(2):254-62. doi: 10.1007/s10461-013-0497-x. PMID 23657758
- [Background] Carballo-Dieguez A, Frasca T, Dolezal C, Balan I. Will gay and bisexually active men at high risk of infection use over-the-counter rapid HIV tests to screen sexual partners? J Sex Res. 2012;49(4):379-87. doi: 10.1080/00224499.2011.647117. Epub 2012 Jan 31. PMID 22293029
- [Background] Thirumurthy H, Masters SH, Mavedzenge SN, Maman S, Omanga E, Agot K. Promoting male partner HIV testing and safer sexual decision making through secondary distribution of self-tests by HIV-negative female sex workers and women receiving antenatal and post-partum care in Kenya: a cohort study. Lancet HIV. 2016 Jun;3(6):e266-74. doi: 10.1016/S2352-3018(16)00041-2. Epub 2016 Apr 8. PMID 27240789
- [Background] Masters SH, Agot K, Obonyo B, Napierala Mavedzenge S, Maman S, Thirumurthy H. Promoting Partner Testing and Couples Testing through Secondary Distribution of HIV Self-Tests: A Randomized Clinical Trial. PLoS Med. 2016 Nov 8;13(11):e1002166. doi: 10.1371/journal.pmed.1002166. eCollection 2016 Nov. PMID 27824882
- [Background] Shannon K, Strathdee SA, Goldenberg SM, Duff P, Mwangi P, Rusakova M, Reza-Paul S, Lau J, Deering K, Pickles MR, Boily MC. Global epidemiology of HIV among female sex workers: influence of structural determinants. Lancet. 2015 Jan 3;385(9962):55-71. doi: 10.1016/S0140-6736(14)60931-4. Epub 2014 Jul 22. PMID 25059947
- [Background] Jakubowski A, Omanga E, Agot K, Thirumurthy H. Large Price Premiums for Unprotected Sex Among Female Sex Workers in Kenya: A Potential Challenge for Behavioral HIV Prevention Interventions. J Acquir Immune Defic Syndr. 2016 May 1;72(1):e20-2. doi: 10.1097/QAI.0000000000000929. No abstract available. PMID 27097367
- [Background] Alary M, Lowndes CM. The central role of clients of female sex workers in the dynamics of heterosexual HIV transmission in sub-Saharan Africa. AIDS. 2004 Apr 9;18(6):945-7. doi: 10.1097/00002030-200404090-00013. No abstract available. PMID 15060443
- [Background] Voeten HA, Egesah OB, Ondiege MY, Varkevisser CM, Habbema JD. Clients of female sex workers in Nyanza province, Kenya: a core group in STD/HIV transmission. Sex Transm Dis. 2002 Aug;29(8):444-52. doi: 10.1097/00007435-200208000-00003. PMID 12172528
- [Background] Skovdal M, Campbell C, Madanhire C, Mupambireyi Z, Nyamukapa C, Gregson S. Masculinity as a barrier to men's use of HIV services in Zimbabwe. Global Health. 2011 May 15;7:13. doi: 10.1186/1744-8603-7-13. PMID 21575149
- [Background] Bwambale FM, Ssali SN, Byaruhanga S, Kalyango JN, Karamagi CA. Voluntary HIV counselling and testing among men in rural western Uganda: implications for HIV prevention. BMC Public Health. 2008 Jul 30;8:263. doi: 10.1186/1471-2458-8-263. PMID 18664301
- [Background] Guidance on Couples HIV Testing and Counselling Including Antiretroviral Therapy for Treatment and Prevention in Serodiscordant Couples: Recommendations for a Public Health Approach. Geneva: World Health Organization; 2012 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK138278/ PMID 23700649
- [Background] Kumwenda M, Munthali A, Phiri M, Mwale D, Gutteberg T, MacPherson E, Theobald S, Corbett L, Desmond N. Factors shaping initial decision-making to self-test amongst cohabiting couples in urban Blantyre, Malawi. AIDS Behav. 2014 Jul;18 Suppl 4(Suppl 4):S396-404. doi: 10.1007/s10461-014-0817-9. PMID 24929834
- [Background] Orasure Techonologies, I., OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test Package Insert. Accessed 14 September 2011 http://www.orasure.com/products-infectious/products-infectious-oraquick.asp: Bethlehem, PA.
- [Background] Bernard, H.R., Research Methods in Anthropology. 1995, Walnut Creek Altamira Press 535.
- [Background] Miles, M.H., A.H., Qualitative Data Analysis: An Expanded Sourcebook, 2nd Edition 1994, Thousand Oaks: Sage Publications
- [Derived] Ruderman LW, Ochwal P, Marcus N, Napierala S, Thirumurthy H, Agot K, Maman S. 'When I have these kits ... I have confidence' - HIV self-testing provides agency for women in their sexual decision-making. Glob Public Health. 2022 Dec;17(12):3735-3746. doi: 10.1080/17441692.2022.2092176. Epub 2022 Jun 30. PMID 35770697
- [Derived] Thirumurthy H, Bair EF, Ochwal P, Marcus N, Putt M, Maman S, Napierala S, Agot K. The effect of providing women sustained access to HIV self-tests on male partner testing, couples testing, and HIV incidence in Kenya: a cluster-randomised trial. Lancet HIV. 2021 Dec;8(12):e736-e746. doi: 10.1016/S2352-3018(21)00248-4. PMID 34856179
- [Derived] Napierala S, Bair EF, Marcus N, Ochwal P, Maman S, Agot K, Thirumurthy H. Male partner testing and sexual behaviour following provision of multiple HIV self-tests to Kenyan women at higher risk of HIV infection in a cluster randomized trial. J Int AIDS Soc. 2020 Jun;23 Suppl 2(Suppl 2):e25515. doi: 10.1002/jia2.25515. PMID 32589354

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Community
Period: Overall Study
Arm/Group | Provision of Multiple Self-tests | Referral Vouchers for VCT
Started | 1063; 33 Community | 1039; 33 Community
Completed | 1019; 33 Community | 991; 33 Community
Not Completed | 44; 0 Community | 48; 0 Community

BASELINE CHARACTERISTICS:
Population: The number of participants at baseline differs from the number of participants in the participant flow: 10 participants were duplicates, thus removed from the study after enrollment; 2 were found to be ineligible after enrollment; 4 participant baseline surveys were lost.
Groups:
- Total: Total of all reporting groups
Arm/Group | Provision of Multiple Self-tests | Referral Vouchers for VCT | Total
Number analyzed (Participants) | 1054 | 1032 | 2086
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [22 to 31] | 25 [22 to 31] | 25 [22 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1054 | 1032 | 2086
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1054 | 1032 | 2086
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 1054 | 1032 | 2086

OUTCOME MEASURES:

1. Primary Outcome: HIV Incidence Per 100 Person Years
Description: HIV incidence over an average follow-up period of 18 months, and up to 24 months, per 100 person years
Time Frame: up to 24 months
Measure: Number; unit: cases per 100 person years
Arm/Group | Provision of Multiple Self-tests | Referral Vouchers for VCT
Number analyzed (Participants) | 1019 | 991
cases per 100 person years | 1.18 | .98

2. Secondary Outcome: Identification of HIV-positive Male Partners
Description: Average number of sexual partners per participant that the participant reported as HIV positive over the course of the study (Total reported positive sexual partners divided by number of participants who completed at least one 6-month follow-up survey); the intent of this measure is to see if participants given HIV self-tests are more likely to identify HIV positive sexual partners.
Time Frame: up to 24 months
Measure: Mean (Standard Deviation); unit: partners per participants
Arm/Group | Provision of Multiple Self-tests | Referral Vouchers for VCT
Number analyzed (Participants) | 1017 | 985
partners per participants | .26 (0.71) | .13 (0.48)

3. Secondary Outcome: Used Condom With at Least One Partner After Partner Refused Self-test or HIV Testing Services Referral Card, or Tested HIV-positive
Description: Percentage of participants who used a condom with at least one sexual partner after partner refused self-test or HIV testing services referral card, or tested HIV-positive; Note that percentages are rounded to one decimal place.
Time Frame: Data was measured longitudinally up to 24 months for some subjects; all participants were measured through 18 months. Measures reported are from 18 month follow-up for behavior occurring in the past 6 months.
Population: Secondary outcomes were assessed at 6, 12, 18, and 24 month surveys. HIV testing (primary outcome) also occurred at 9, 15, and 21 months, so the number of overall participants may not match what is reported for the primary outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Provision of Multiple Self-tests | Referral Vouchers for VCT
Number analyzed (Participants) | 1017 | 985
percentage of participants
  6 months: number analyzed (Participants) | 921 | 915
  6 months | 11.6 | 6.2
  12 months: number analyzed (Participants) | 898 | 887
  12 months | 7.2 | 5.2
  18 months: number analyzed (Participants) | 949 | 891
  18 months | 5.3 | 4.3
  24 months: number analyzed (Participants) | 302 | 268
  24 months | 3.3 | 4.9

4. Secondary Outcome: Couples Testing With Primary Partner
Description: Percentage of participants who report testing together with their primary partner; Note that percentages are rounded to one decimal place.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Provision of Multiple Self-tests | Referral Vouchers for VCT
Number analyzed (Participants) | 1017 | 985
percentage of participants
  6 months: number analyzed (Participants) | 921 | 915
  6 months | 80.3 | 32.9
  12 months: number analyzed (Participants) | 898 | 887
  12 months | 75.3 | 34.7
  18 months: number analyzed (Participants) | 949 | 891
  18 months | 34.7 | 26.7
  24 months: number analyzed (Participants) | 302 | 268
  24 months | 71.6 | 26.2

5. Secondary Outcome: Primary Partner Tested for HIV
Description: Percentage of participants who report that their primary partner tested for HIV since enrollment; Note that percentages are rounded to one decimal place.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Provision of Multiple Self-tests | Referral Vouchers for VCT
Number analyzed (Participants) | 1017 | 985
percentage of participants
  6 months: number analyzed (Participants) | 921 | 915
  6 months | 87.5 | 48.3
  12 months: number analyzed (Participants) | 898 | 887
  12 months | 81.2 | 48.6
  18 months: number analyzed (Participants) | 949 | 891
  18 months | 77.8 | 39.8
  24 months: number analyzed (Participants) | 302 | 268
  24 months | 74.9 | 39

6. Secondary Outcome: Declined Sex With at Least One Partner After Partner Refused Self-test or HIV Testing Services Referral Card, or Tested HIV-positive
Description: Percentage of participants who declined sex with at least one partner after partner refused self-test or HIV testing services referral card, or tested HIV-positive; Note that percentages are rounded to one decimal place.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Provision of Multiple Self-tests | Referral Vouchers for VCT
Number analyzed (Participants) | 1017 | 985
percentage of participants
  6 months: number analyzed (Participants) | 921 | 915
  6 months | 14.2 | 7.1
  12 months: number analyzed (Participants) | 898 | 887
  12 months | 5.1 | 6
  18 months: number analyzed (Participants) | 949 | 891
  18 months | 4.5 | 3.8
  24 months: number analyzed (Participants) | 302 | 268
  24 months | 2.3 | 3

7. Other Pre Specified Outcome: Intimate Partner Violence (IPV)
Description: Percentage of participants in each study group who experience IPV; Note that percentages are rounded to one decimal place.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Provision of Multiple Self-tests | Referral Vouchers for VCT
Number analyzed (Participants) | 1017 | 985
percentage of participants
  6 months: number analyzed (Participants) | 921 | 915
  6 months | 17.3 | 16.4
  12 months: number analyzed (Participants) | 898 | 887
  12 months | 10.8 | 17.7
  18 months: number analyzed (Participants) | 949 | 891
  18 months | 6.1 | 3.5
  24 months: number analyzed (Participants) | 302 | 268
  24 months | 5.0 | 5.2

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and recorded for the full 24 month duration of the study (June 4, 2017 - March 25, 2020).
Description: Other (Not Including Serious) Adverse Events for this study was categorized as Intimate partner violence (IPV) and social harms. IPV was only assessed via 6-month surveys, so the denominators vary from other AE categories.
Arm/Group | Provision of Multiple Self-tests | Referral Vouchers for VCT
All-Cause Mortality (participants affected / at risk) | 1/1019 | 1/991
Serious Adverse Events (participants affected / at risk) | 0/1019 | 0/991
Other Adverse Events (participants affected / at risk) | 241/1017 | 210/985
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Provision of Multiple Self-tests (N=1017) | Referral Vouchers for VCT (N=985)
Intimate partner violence and social harms (Social circumstances) | 241 | 210 — Individuals who reported ever experiencing intimate partner violence (IPV) while participating in the study, that may or may not have been related to study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT03135067/Prot_SAP_000.pdf